CLINICAL TRIAL: NCT03580564
Title: An Open, Multicenter Phase II Study to Evaluate the Safety and Efficacy of KL-A167 Injection in Relapsed or Refractory Classical Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KL167-Ⅱ-03-CTP
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — 18-O-demethylcervinomycin A2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): KL-A167 900 mg intravenously (IV) every-2-weeks (Q2W)
  Interventions: Drug: KL-A167

INTERVENTIONS:
Drug: KL-A167 — KL-A167 900 mg intravenously (IV) every-2-weeks (Q2W)

SUMMARY:
The study is to evaluate the efficacy of KL-A167 a in subjects with relapsed or refractory classical Hodgkin lymphoma (cHL), as measured by Overall Response Rate (ORR) per the Lugano Classification

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Histopathological confirmed classical Hodgkin's lymphoma
* Relapsed/refractory cHL include：subject with no response to or with progression after ASCT ；subject which failed failed second line and above chemtherapy；subject which didn't achieve PR after 2 cycles or didn't achieve CR after 4 cycles
* At least one measurable disease (long axis>15 mm and short axis>5 mm,or both axis>10 mm）
* ECOG performance status of 0 or 12
* Subject must have adequate organ functions and meet requirements on laboratory values.：Count of Blood Cells: absolute neutrophil count (ANC) ≥ 1.0 × 109 / L; platelet count (PLT) ≥ 50 × 109 / L; hemoglobin content (HGB) ≥ 7.0 g / Dl; Liver function: serum total bilirubin (TBIL) ≤ 1.5 × normal upper limit (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN，with the exception of patients with hepatic metastases (ALT and AST ≤ 5 × ULN) and patients with hepatic metastases or Gilbert's syndrome (total bilirubin ≤ 3 × ULN)Renal function: serum creatinine (Cr) ≤ 1.5 × ULN or Creatinine clearance rate（CCR）≥50 mL/min；International normalized ratio (INR) ≤ 1.5 x ULN ；Thyroid function: thyroid stimulating hormone (TSH) in normal range.
* Prior chemotherapy, radiotherapy, immunotherapy or investigational therapy (including Chinese herbal medicine and Chinese patent medicine) used to control cancer including locoregional treatment must have been completed ≥ 4 weeks before the first dose of KL-A167(Mitomycin or nitroso must have been completed ≥ 6 weeks), and all treatment-related adverse events (except alopecia) are stable and have either returned to baseline or Grade 0/1
* Subjects of reproductive potential must be willing to use adequate contraception during the course of the study and through 6 months after the last dose of study medication
* Subject has voluntarily agreed to participate by giving written informed consent.

Exclusion Criteria:

* Nodular lymphocyte-predominant Hodgkin lymphoma or gray zone lymphoma.
* Known central nervous system lymphoma.
* Prior malignancy except for curatively treated carcinoma in situ of the cervix or breast ，Superficial bladder cancer，and Squamous cell carcinoma in situ
* History of severe hypersensitivity reaction to monoclonal antibodies
* Prior exposure to any anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibody.
* need the other anticancer therapy during the study
* Received any anticancer vaccine or other medications for immunomodulatory receptor preparations
* Received HSCT
* Received ASCT in the past 3 months
* Serious acute or chronic infection requiring systemic therapy.
* Subject with active autoimmune disease or history of autoimmune disease with high risk of recurrence.
* Conditions requiring systemic treatment with either corticosteroids (> 10 mg daily Prednisone equivalent) or other immunosuppressive medications within 14 days of first dose of KL-A167
* serious medical diseases, ex Suffering from heart failure (New York Heart Association standard III or IV), ischemic heart disease (such as myocardial infarction or angina), congestive heart failure and other cardiovascular diseases, uncontrolled diabetes(fasting blood glucose≥10 mmol/L), uncontrolled high blood pressure(Systolic> 150 mmHg and / or diastolic> 100 mmHg), LVEF<50%
* QTcF>450 msec
* Known active HBV or HCV infection.
* Known HIV infection.
* Has history of interstitial lung disease or non-infectious pneumonitis. Subjects with prior drug-induced or radiation-induced pneumonitis who are asymptomatic are eligible.
* Known active pulmonary tuberculosis
* Has history of AE related with immune system during the Immunotherapy
* Received a live vaccine within 4 weeks of the first dose of study medication or plan to receive live vaccine during study period.
* Known neurological or psychiatric diseases
* Ongoing alcohol or drug abuse
* Pregnancy (absence to be confirmed by serum β-human chorionic gonadotropin test) or breastfeeding
* Participation in another clinical trial within the past 4 weeks
* Other significant disease that in the investigator's opinion should exclude the subject from the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-08-22 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 2years
  Overall Response Rate (ORR) defined as the proportion of subjects who achieves a best response of CR or PR, assessed by IRC per the Lugano Classification

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to 2years
  From the first dose of KL-A167 to the date of PD or death, whichever occurs first
Duration of Response (DOR) | Up to 2years
  From the date that response criteria are first met to the date that PD is objectively documented or death, whichever occurs first
Overall Survival (OS) | Up to 2years
  From the first dose of KL-A167 to the date of death
Time to Response | Up to 2years
  From the date of the first dose of KL-A167 to the time the response criteria are first met

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China